CLINICAL TRIAL: NCT00504712
Title: A Randomised, Double Blind, Placebo Controlled, Parallel Pilot Study to Test the Effect of Testosterone Treatment on Peripheral Vascular Disease in Hypogonadal Men With Type 2 Diabetes Mellitus
Brief Title: Testosterone for Peripheral Vascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barnsley Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 300
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2022-05-18 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-03

CONDITIONS: Hypogonadism; Peripheral Vascular Disease; Type 2 Diabetes
Keywords: Testosterone; Hypogonadism; Diabetes; PVD; RCT
MeSH Terms: conditions — Hypogonadism; Peripheral Vascular Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Testosterone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Testosterone 200 mg intramuscular every 2 weeks
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Testosterone — Sustanon- 200mg- Intramuscular testosterone every 2 weeks
  Arms: Active
Drug: saline — Saline injection every two weeks
  Arms: Placebo

SUMMARY:
There is increasing evidence of the linkage of type 2 diabetes with low testosterone levels in men.

DETAILED DESCRIPTION:
Testosterone treatment has shown beneficial effects on blood sugar control and obesity in pilot studies in men with type 2 diabetes. Beneficial effects have also been seen on angina- a disease related to atherosclerosis (narrowing of the arterial blood vessels). Peripheral vascular disease is also caused by atherosclerosis. We hypothesise that testosterone will have beneficial effects on peripheral vascualr disease in men with low serum testosterone and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus.
2. Serum testosterone 12 nmol/L or less on two consecutive samples taken on different days and symptoms compatible with hypogonadism.
3. Peripheral vascular disease as defined by

   * previous diagnosis by a specialist vascular surgeon OR
   * ABPI less than 0.92 and ischaemic leg pain (claudication or rest pain) or distal complications (non-healing arterial foot ulcer or gangrene).
4. Agreement to maintain antihypertensive and antilipid treatments at prior doses during 3 month duration of study.
5. Ability to give written informed consent after verbal and written explanation in the English language.
6. Ability to comply with all study requirements.

Exclusion Criteria:

1. Current or previous breast cancer.
2. Current or previous prostate cancer.
3. Raised prostate specific antigen (PSA) or abnormal per rectal examination unless prostate cancer excluded after specialist urology opinion.
4. Severe symptoms of benign prostatic hypertrophy ('prostatism')
5. Treatment with testosterone in the 3 months prior to the trial.
6. Investigational drug treatment in the 3 months prior to the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Jones, Principal Investigator — Barnsley Hospital
Locations (1):
- Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: started 02/02/2006
Period: Overall Study
Arm/Group | Active | Placebo
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants were men aged greater than 40 years
  years | 56.6 (11.9) | 61.7 (11.8) | 59.15 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 13 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Arterial Stiffness
Description: The primary outcome was the effect of 12 weeks testosterone replacement on arterial stiffness measured by ultrasound derived stiffness parameter β of the femoral artery. A reduction in ultrasound derived stiffness parameter β is clinically beneficial to patients and the study was looking for a reduction in this value. Stiffness index β was calculated from the diastolic carotid artery diameter (Dd), systolic carotid artery diameter (Ds), diastolic blood pressure (BPd) and systolic blood pressure (BPs) using the formula; Stiffness index β = (ln(Ps/Pd)) x Dd/(Ds-Dd). A full theoretical range of possible index scores does not exist.
Time Frame: Baseline, 12 weeks, and 26 weeks
Measure: Mean (Standard Deviation); unit: index β
Arm/Group | Active | Placebo
Number analyzed (Participants) | 11 | 13
index β
  Baseline | 15.02 (5.74) | 15.08 (6.59)
  12 weeks | 14.08 (5.36) | 16.12 (7.42)
  26 weeks | 14.01 (4.53) | 12.58 (5.55)

2. Secondary Outcome: Change in IMT
Description: Progression of Carotid intima-media thickness measured in mm
Time Frame: Baseline, 12 weeks, and 26 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active | Placebo
Number analyzed (Participants) | 11 | 13
mm
  Baseline | 0.856 (0.132) | 0.885 (0.130)
  12 weeks | 0.843 (0.137) | 0.887 (0.120)
  26 weeks | 0.841 (0.135) | 0.872 (0.124)

ADVERSE EVENTS:
Description: Specific Adverse Event terms were not used for this study.
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/13
Other Adverse Events (participants affected / at risk) | 3/11 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=11) | Placebo (N=13)
Serious (Cardiac disorders) | 1 (1) | 0 (0) — Admitted with chest pain and shortness of breath. Diagnosis was obstructive sleep apnoea and exacerbation of known heart failure
Serious (General disorders) | 0 (0) | 1 (1) — Admitted with worsening foot ulceration, heart failure and acute kidney injury
Adverse Event (Renal and urinary disorders) | 0 (0) | 1 (1) — Diagnosed bladder cancer
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=11) | Placebo (N=13)
Adverse Event (General disorders) | 1 (1) | 0 (0) — viral illness
Adverse (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — chest infection
Adverse (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — post injection muscle haematoma
Adverse (General disorders) | 0 (0) | 1 (1) — fracture of humerus,
Adverse (General disorders) | 0 (0) | 1 (1) — unilateral calf swelling with no DVT
adverse (Infections and infestations) | 0 (0) | 1 (1) — viral infection
Adverse (General disorders) | 0 (0) | 1 (1) — gynaecomastia

LIMITATIONS AND CAVEATS:
It was more difficult than anticipated to recruit patients to the trial and despite extension of the trial beyond expected completion date the target recruitment was not achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes